CLINICAL TRIAL: NCT02815449
Title: Assessment of the Bioavailability of Iron in Iron Fortified Bouillon Cubes in Healthy Nigerian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Obafemi Awolowo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: FDS-SAV-2103
Record Dates: First submitted 2016-05-24; First posted 2016-06-28 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron fortification; Bioavailability; Nigeria; Women; Bouillon cubes
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low stabilizer level (Experimental): Meals prepared with iron fortified cube with low stabilizer level
  Interventions: Other: Meals prepared with iron fortified cube with Low stabilizer level
- Medium stabilizer level (Experimental): Meals prepared with iron fortified cube with medium stabilizer level
  Interventions: Other: Meals prepared with iron fortified cube with Medium stabilizer level
- High stabilizer level (Experimental): Meals prepared with iron fortified cube with high stabilizer level
  Interventions: Other: Meals prepared with iron fortified cube with High stabilizer level

INTERVENTIONS:
Other: Meals prepared with iron fortified cube with Low stabilizer level — Meals prepared with iron fortified cube with Low stabilizer level
  Arms: Low stabilizer level
Other: Meals prepared with iron fortified cube with Medium stabilizer level — Meals prepared with iron fortified cube with Medium stabilizer level
  Arms: Medium stabilizer level
Other: Meals prepared with iron fortified cube with High stabilizer level — Meals prepared with iron fortified cube with High stabilizer level
  Arms: High stabilizer level

SUMMARY:
The prevalence of iron deficiency anemia is a wide spread problem in Africa and iron fortification can be an effective strategy to decrease this.

In the current study adding different levels of a stabilizer to iron fortified cubes and it's effect on iron bioavailability from these cubes will be studied in the context of a Nigerian meal in women.

24 Female subjects with low serum ferritin levels will be included in the study. The study will last 64 days and subjects will be asked to consume a breakfast and lunch prepared with a bouillon cube with isotope labeled iron during 3 periods of 5 consecutive days. The absorption of iron will be evaluated after every period and compared between the cubes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female Nigerian subjects;
* Age > 18 and <40 years at screening;
* Body weight <65 kg;
* Apparently healthy: no medical conditions which might affect study measurements (judged by study physician);
* With iron deficiency judged by a serum ferritin concentration of <15µg/L;
* Reported intense sporting activities ≤ 10h/w;
* Reported alcohol consumption ≤ 14 units/w;
* Willing and able to participate in the study;
* Having given a written informed consent.

Exclusion Criteria:

* Being an employee of Unilever or the Department of Family, Nutrition and Consumer Science of the Obafemi Alowolo University;
* Blood donation or significant blood loss over the past 6 months;
* Being severely anemic (hemoglobin < 8.0 g/dL)
* Reported use of any medically- or self-prescribed diet;
* Use of vitamin or mineral supplements and unwillingness to discontinue their use one week prior the study and during the study;
* Smoking or consuming tobacco in any form, and/or was smoking or consuming tobacco in any form for 6 months preceding the study and/or will be smoking or consuming tobacco in any form, during the study;
* Is pregnant or will be planning pregnancy during the study period;
* Is lactating or has been lactating in the 6 weeks before pre-study investigation and/or during the study period;
* Known gastrointestinal (including helminth infection) or metabolic disorders;
* Participation in another clinical trial during the last 30 days prior to the beginning of the study;
* Symptomatic malaria (no blood smear analyses on malaria required)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Iron isotopic composition of the blood at the end of each intervention period | 16 days
  The amount of iron isotopic label in the blood will be related to the low, medium and high stabilizer level in the cubes to determine whether a dose-response relationship exists.

SECONDARY OUTCOMES:
Iron isotopic composition of the blood | 1, 22, 43 and 64 days
  The amount of iron isotopic label in the blood at the end of each administration period plus 14 day incorporation time will be used to calculate the absolute Iron absorption for each stabilizer level

CONTACTS AND LOCATIONS:
Overall Officials: Funke Olumakaiye, PhD, Principal Investigator — Obafemi Awolowo University
Locations (1):
- Obafemi Owalowo University, Ile-Ife, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eilander A, Funke OM, Moretti D, Zimmermann MB, Owojuyigbe TO, Blonk C, Murray P, Duchateau GS. High Bioavailability from Ferric Pyrophosphate-Fortified Bouillon Cubes in Meals is Not Increased by Sodium Pyrophosphate: a Stable Iron Isotope Study in Young Nigerian Women. J Nutr. 2019 May 1;149(5):723-729. doi: 10.1093/jn/nxz003. PMID 31004134